CLINICAL TRIAL: NCT05190835
Title: Quantification and Characterization of Foot Postoperative Edema - Bicentric Prospective Study
Brief Title: Quantification and Characterization of Foot Postoperative Edema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique MEGIVAL (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-A01802-39
Record Dates: First submitted 2021-12-10; First posted 2022-01-13 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Surgery--Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hallux surgery (Other): These are patients operated on for hallux without change of strategy compared to current care
  Interventions: Device: Optical scanner
- Metatarsal paddle surgery (Other): These are patients operated on for metatarsal paddle without change of strategy compared to current care
  Interventions: Device: Optical scanner
- Hallux and metatarsal pallet surgery (Other): These are patients operated on for hallux and metatarsal paddle without change of strategy compared to current care
  Interventions: Device: Optical scanner

INTERVENTIONS:
Device: Optical scanner — During the visits (Day 0 before surgery, Day 8, Day 21, Day 45, Month 3 and Month 6 after surgery), a measurement of the volume and the perimeter of the patient's two feet is carried out (operated foot and control foot). The edema is measured by a non-invasive method using an optical scanner (camera + laser scanning). The image processing software accompanying this tool has an automatic calculation of the volumes and the different perimeters of the foot. The measurement time by the scanner is less than 4 seconds.

SUMMARY:
In foot surgery, postoperative edema is a complication making the postoperative outcome quite uncertain as to the rehabilitation of the patient. The evolution of this edema is unknown ... The means of "mastering" this edema are empirical, with little study other than cryotherapy and restraint. This study aims to study postoperative edema in a cohort of patients undergoing forefoot surgery. The follow-up will be prospective with measurement of the volume of the foot using an optical technique, during the various follow-up consultations between Day 8 and Month 6 postoperative.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Patient operated on forefoot surgery
* Patient having given informed consent
* For female patients of childbearing age, not to be pregnant or likely to be during the study, not to be breastfeeding

Exclusion Criteria:

* Minor patient
* Patient deprived of his liberty or under guardianship
* Patient operated on for surgery of the forefoot other than hallux and lateral toes
* Patient unable to undergo protocol monitoring for psychological, social, family, geographic or linguistic reasons
* Patient with an underlying or concomitant pathology incompatible with inclusion in the trial, whether psychiatric or somatic
* Vulnerable people according to article L1121-6 of the CSP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Evaluate the change of volume of an operated foot to evaluate the edema. | Day 0 before surgery, Day 8 after surgery
  Change of volume of the foot from Day 0
Evaluate the change of volume of the edema of an operated foot during the 6 months after surgery | Day 21, Day 45, Month 3 and Month 6 after surgery

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Polyclinique Saint Roch, Montpellier
  - Clinique MEGIVAL, Saint-Aubin-sur-Scie

IPD SHARING:
Plan to Share IPD: Undecided